CLINICAL TRIAL: NCT01337609
Title: A Double-Blind, Placebo-Controlled Study of the Probiotic Ganeden BC30 (Bacillus Coagulans GBI-30, 6068) in Irritable Bowel Syndrome Comorbid With Major Depressive Disorder (MDD)
Brief Title: Study of Probiotic GanedenBC30 for Irritable Bowel Syndrome and Major Depressive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because the study sponsor chose to discontinue funding for this protocol following a change in leadership, the study was terminated early.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ganeden Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008P002387
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder; Irritable Bowel Syndrome
Keywords: Depression; Irritable Bowel Syndrome; Probiotic; Bacillus Coagulans
MeSH Terms: conditions — Depressive Disorder, Major; Irritable Bowel Syndrome; Depression | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GanedenBC30 (Experimental): Arm 1 will take GanedenBC30 (Bacillus coagulans GBI-30, 6086, 1 capsule/day) for 60 days.
  Interventions: Drug: Ganeden BC30
- Sugar pill (Placebo Comparator): Arm 2 will take placebo (sugar pill) for 60 days.
  Interventions: Other: Placebo (sugar pill)
- Ganeden BC30, Sugar pill (Other): Arm 3 will take placebo (sugar pill) for 30 days, followed by Ganeden BC30 for 30 days.
  Interventions: Other: Ganeden BC30, Placebo (sugar pill)

INTERVENTIONS:
Drug: Ganeden BC30 — 2 billion CFU per capsule; One pill daily for 60 days
  Arms: GanedenBC30
Other: Placebo (sugar pill) — 1 pill daily for 60 days
  Arms: Sugar pill
Other: Ganeden BC30, Placebo (sugar pill) — Ganeden BC30 (2 billion CFU per capsule), One capsule daily for 30 days Sugar Pill (placebo), One capsule daily for 30 days
  Arms: Ganeden BC30, Sugar pill

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a nutritional supplement, the probiotic bacteria GanedenBC30. Probiotics are live microorganisms which when taken in large enough amounts are supposed to provide a health benefit. The investigators would like to see whether this supplement can be used as a treatment for Irritable Bowel Syndrome (IBS) and Major Depressive Disorder (MDD). Participants in the study will have both IBS and MDD. In order to find out if GanedenBC30 is effective in treating IBS and MDD, the investigators will compare it to a placebo. About 32 people will take part in this research study. About half of these 32 people will take part at Charles River Medical Associates and half will take part at Burlington Medical Associates. Participants will be recruited from among patients already being seen at Charles River Medical Associates or Burlington Medical Associates for their primary care. The study will last for two months, during which time participants will make eight study visits and will take either Ganeden BC30 or placebo. The investigators hypothesize that subjects treated with the probiotic will have significantly better outcomes with regard to depression and IBS symptoms compared to those who receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Able to give Informed Consent
* Meet criteria for Irritable Bowel Syndrome
* Meet criteria for Major Depressive Disorder
* Men and women ages 18 to 65
* Women of childbearing potential must be using an adequate methods of contraception
* Can be on an antidepressant medications, but must have been on the medication for at least 8 weeks and at a stable dose for 4 weeks
* Can be on medications for IBS, but must have been on medications for at least 8 weeks and at a stable dose for 4 weeks

Exclusion Criteria:

* Patients who have failed one or more trials of probiotics for IBS
* Patients who report an inadequate response to less than two or more than four adequate trails of antidepressant treatments during the current depressive episode at a therapeutic dose for an adequate duration
* Women who are pregnant or breastfeeding
* Patients with "alarm signs" or "red flags" as defined by American Gastroenterological Association (AGA) are excluded [6], unless they have been fully evaluated to rule out other significant diseases.
* Patients with known diagnoses of digestive organic disease, celiac disease and lactose intolerance prior to the screening.
* Patients who report an inadequate response (less than 50% decrease in depressive symptom severity) to less than two or more than four prior adequate trials of antidepressant treatments during the current depressive episode (including monotherapy treatment and distinct combination regimens) at a therapeutic dose (as defined by the MGH-ATRQ) and for an adequate duration (minimum six weeks for any monotherapy).
* Patients who report treatment with adjunctive medications to their antidepressant for a minimum of four weeks during the current depressive episode.
* Patients with a current need for involuntary commitment or who have been hospitalized within four weeks of the Screening Visit for the current major depressive episode.
* Patients who have received ECT during the current episode.
* Patients who have a current Axis I diagnosis of:

Delirium, dementia, amnestic, or other cognitive disorder; Schizophrenia or other psychotic disorder, based on the PDSQ; Bipolar I or II disorder, based on the PDSQ; Patients with a clinically significant Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.

* Patients experiencing hallucinations, delusions, or any psychotic symptomatology in the current depressive episode.
* Patients who have met DSM-IV-TR criteria for any significant substance use disorder within the past six months, based on the PDSQ.
* Patients receiving new onset depression-focused psychotherapy within 6 weeks of screening, or at any time during participation in the trial.
* Patients who have been previously randomized in a probiotics clinical trial (lifetime).
* Patients who have participated in any clinical trial with an investigational drug or device within the past month.
* Patients who, in the opinion of the investigator, are actively suicidal or homicidal and at significant risk for suicide or homicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Burlington Medical Associates, Burlington, Massachusetts
  - Charles River Medical Associates, Westborough, Massachusetts

REFERENCES:
- See also: Massachusetts General Hospital Depression Clinical and Research Program Website — http://massgeneral.org/depression

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Started | 1 | 2 | 2
Completed | 0 | 2 | 2
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill | Total
Number analyzed (Participants) | 1 | 2 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Description: The Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)is a self report measure that addresses depressive symptoms. MDD responders will be defined as those exhibiting a 50% decrease in the QIDS SR at study endpoint.
Time Frame: Administered at each of 8 study visits (every 10 days), Endpoint is Final Visit
Population: Because the study sponsor chose to discontinue funding for this protocol following a change in leadership, the study was terminated early and this outcome measure was not analyzed.
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: IBS Severity Scoring System (IBS-SSS)
Description: The IBS-SSS is a validated instrument used to assess common IBS symptoms over the past 10 days including abdominal pain, distention, bowel habit, and global function. The IBS-SSS will be used to assess the absolute change in specific IBS symptoms at endpoint, namely the bloating/distension score.
Time Frame: Adminsitered at each of 8 study visits (every 10 days), Endpoint is Final Visit
Population: as for outcome 1
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Visual Analog Scale (VAS)
Description: The VAS is a self-administered measure of abdominal pain, discomfort, and bloating. The change in total score from baseline to study endpoint will be assessed.
Time Frame: Administered at each of 8 study visits (every 10 days), Endpoint is Final Visit
Population: as for outcome 1
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Adequate Relief of IBS Pain (AR-IBS)
Description: The AR-IBS is a self-administered measure of the adequacy of the relief of IBS pain.
Time Frame: Adminstered at each of 8 visits (every 10 days), Endpoint is Final Visit
Population: as for outcome 1
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Patient Global Impression of Change (PGI-C) - IBS Symptoms
Description: The PGI-C is a self-administered measure of the degree of improvement in IBS symptoms compared to the first study visit. Degree of improvement in IBS symptoms from first to final visit will be assessed using this scale.
Time Frame: Administered at each of 8 visits (every 10 days), Endpoint is Final Visit
Population: as for outcome 1
Arm/Group | GanedenBC30 | Sugar Pill | Ganeden BC30, Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo for 60 Days | GanedenBC30 for 60 Days | Placebo for 30 Days, Followed by GanedenBC30 for 30 Days
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/1 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo for 60 Days (N=2) | GanedenBC30 for 60 Days (N=1) | Placebo for 30 Days, Followed by GanedenBC30 for 30 Days (N=2)
Cerebral infarct; residual leg weakness and face drooping (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study treatment
Labial cyst, constipation, and tension headache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study treatment
Sore throat (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study treatment
Sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study treatment
Right flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study treatment

LIMITATIONS AND CAVEATS:
Because the study sponsor chose to discontinue funding for this protocol following a change in leadership, the study was terminated early and data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No